CLINICAL TRIAL: NCT05970575
Title: Open Label Phase IIa Study Evaluating the Safety and Efficacy of NE3107 in Improving Sleep and Fatigue in Subjects With Traumatic Brain Injury
Brief Title: Insulin-sensitizing NE3107 in Improving Sleep and Fatigue in Subjects With Traumatic Brain Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study team was informed by the final participant's PCP that the subject discontinued the study medication. The participant's caregiver requested for the participant to be withdrawn from the study. The investigator has decided to close out.
Sponsor: Neurological Associates of West Los Angeles (Other)
Collaborators: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NE3107-TBI-TRP
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm: NE3107 (Experimental): All participants will take 200mg BID (12 hours apart) of NE3107 for 6 months.
  Interventions: Drug: NE3107

INTERVENTIONS:
Drug: NE3107 — Participants will take 20mg twice daily (BID) approximately 12 hours apart. The dose will be stable the duration of the study intervention (6 months)

SUMMARY:
This study seeks to measure changes in cognition through verbal and visual test procedures and changes in biomarkers of Traumatic Brain Injury and inflammatory and metabolic parameters.

DETAILED DESCRIPTION:
A growing body of literature recognizes neuroinflammation as a pivotal contributor to the pathogenesis of TBI. A surge of inflammatory cytokines and chemokines, including tumor necrosis factor-alpha (TNF-α), interleukin-1 (IL-1), interleukin-6 (IL-6), and nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB), often follows TBI, leading to a complex cascade of secondary events that ultimately result in neuronal damage and long-term consequences.

It has been shown that patients with mild TBI have higher plasma inflammatory cytokine levels than those without TBI at both 24 hours and 6 months following initial injury.The activation of these inflammatory mediators has been demonstrated in both cerebrospinal fluid (CSF) and serum of TBI patients. Elevated levels of TNF-α in CSF and serum have been associated with injury severity and unfavorable outcomes in TBI.

IL-1, IL-6, and TNF-α induce the extracellular signal-regulated kinase (ERK) pathway, promoting neuroinflammation. Furthermore, NF-kB, a crucial transcription factor in the inflammatory response, plays a significant role in amplifying neuroinflammation post-TBI, mediating the expression of several inflammatory cytokines and contributing to neuronal apoptosis and cognitive impairment.

Neuroinflammation's contribution to sleep disturbances, fatigue, and cognitive impairment has been increasingly recognized. These inflammatory cytokines may influence the hypothalamic-pituitary-adrenal (HPA) axis and disrupt sleep architecture, leading to sleep disturbances and fatigue. Further, they are known to induce synaptic alterations and neuronal apoptosis, contributing to cognitive impairment.

Chronic, low-grade inflammation often ensues post-TBI, contributing to the persistent and potentially insidious process leading to long-term impairment and diminished quality of life.

Apart from neuroinflammation, intracranial insulin resistance, another secondary consequence of TBI, plays a significant role in the pathogenesis of TBI. Insulin resistance has been observed in TBI patients, and it's linked to worse outcomes. In mouse models, induced TBI has been shown to demonstrate reduced glucose uptake in mice brains on positron emission tomography (PET) scans, consistent with the insulin resistance that has been seen in TBI patients. Insulin resistance may exacerbate neuroinflammation, disrupt synaptic plasticity, and contribute to cognitive deficits, further compounding the injury's impact.

If these symptoms remain untreated, they can significantly impair quality of life, limiting independent living and reducing the ability to perform daily activities. They can also predispose individuals to mental health disorders such as depression and anxiety and lead to a higher risk of chronic diseases and premature death.

Currently, there is no therapeutic option to halt or fully reverse the sequelae from traumatic brain injuries or the attendant neurophysiological deterioration. Other conditions with similarly limited-to-no available and effective treatment strategies, including Alzheimer's disease, share an overlapping deteriorative quality relating to neuroinflammation and even reduced insulin functioning. A promising area of research among traumatic brain injury and Alzheimer's treatment is investigating the use of insulin synthesizers; this study group has also initiated a project involving NE3107 among patients with Alzheimer's disease (IND 159271). In addition to IND 159271, several Phase 3 studies had been previously initiated and/or completed with compounds such as Semaglutide, a hormone that stimulates insulin signaling, Metformin, an insulin synthesizer , and NE3107, an anti-inflammatory insulin-sensitizing agent.

In this study, the drug under investigation is NE3107 (17a-ethynyl0androst-5-ene-3b, 7b, 17b-triol). NE3107 is a small, blood-brain permeable molecule with anti-inflammatory and insulin-sensitizing properties. The mechanism of action for NE3107 involves selective inhibition of inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of traumatic brain injury, confirmed by neurologist or other medical professional

Age within range of 18-75 years old

Multidimensional Fatigue Inventory (MFI) score of 27 or greater

Epworth Sleepiness Scale (ESS) score of 10 or greater AND/OR a Pittsburgh Sleep Index (PSI) score of 5 or greater

Ability to Consent: Participants need to be capable of giving informed consent or have a legally authorized representative who can do so.

Ability to participate for the duration of the study

Exclusion Criteria:

* In order for a subject to be considered for this study, he/she may NOT have any of the following:

Diagnosis of other chronic Neurological Conditions: Examples are participants with other pre-existing neurological conditions, such as Alzheimer's or Parkinson's Disease or untreated epilepsy.

Severe Psychiatric Illness: Conditions such as schizophrenia, bipolar disorder, or severe depression.

Current diagnosis of Substance Abuse Disorder, including opioid use disorder.

Dysphagia or Significant GI dysmotility or conditions that would significantly impair absorption

Significant language impairment with expressive or receptive aphasia

Hematological or Metabolic derangement or diagnosis of other medical condition that could be negatively affected by participating in this clinical trial.

Pregnant or plans for pregnancy or breastfeeding during the course of the study

Diagnosis of genetic or developmental disorder with cognitive impairment

Use of more than 2 sleep aids including melatonin

Advanced stages of any terminal illness or any active cancer that requires chemotherapy

History of breast cancer

Women with child-bearing potential who are not willing to use a double-barrier birth control method

Males not willing to use a double-barrier birth control method with female sex partners with child-bearing potential

Individuals with hepatic impairment as defined by:

Alanine aminotransferase (ALT) lab values >3x the upper normal limit (UNL)

Aspartate aminotransferase (AST) lab values >3x UNL

OR

History of clinically significant liver disease in the Principal Investigator's medical judgment

Individuals with renal impairment as defined by Creatinine clearance (Cockcroft-Gault formula) of <45 mL/min.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Safety as Assessed by Quantification of Adverse Events | up to 6 months
  Primary outcome will be collection of AEs and SAEs
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 3 months, 6 months
  a tool used to measure the quality and patterns of sleep
Multidimensional Fatigue Inventory (MFI) | Baseline, 3 Months, 6 Months
  to measure overall fatigue

SECONDARY OUTCOMES:
Montreal Objective Cognitive Assessment change | Baseline, 3 Months, 6 Months
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.

CONTACTS AND LOCATIONS:
Locations (1):
- The Regenesis Project, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No